CLINICAL TRIAL: NCT03196076
Title: Contrast-enhanced Ultrasound for Complex Kidney Lesion Diagnosis in Patients With CKD Extension (CEUS CKDx)
Brief Title: Contrast-enhanced Ultrasound for Complex Kidney Lesion Diagnosis in Patients With CKD Extension
Acronym: CEUS-CKDx
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Lantheus Medical Imaging (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-1130
Record Dates: First submitted 2017-06-20; First posted 2017-06-22 (Actual); Results first posted 2021-07-15 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-06

CONDITIONS: Chronic Kidney Diseases; Cystic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Diseases, Cystic | interventions — perflutren

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Perflutren Lipid Microsphere (Healthy subjects) (Experimental): Healthy subjects will be imaged using contrast-enhanced ultrasound (perflutren) for image optimization prior to enrolling clinical patients.
  Interventions: Drug: Perflutren Lipid microsphere
- Perflutren Lipid Microsphere (patients with kidney lesions) (Experimental): Patients with kidney lesions will be imaged using contrast-enhanced ultrasound with perflutren.
  Interventions: Drug: Perflutren Lipid microsphere
- Controls: No interaction (No Intervention): Patients with kidney lesions will be included as control subjects. These patients will be followed, but will not receive any study intervention.

INTERVENTIONS:
Drug: Perflutren Lipid microsphere — Perflutren will be administered in a bolus or continuous infusion using the dosing range and administration type within the perflutren prescribing information.Once perflutren lipid has been administered, the transducer is maintained in a constant position over the area of interest to show the target lesion in order to assess the enhancement pattern during the early, mid and late vascular phases. Images will also be taken of kidney parenchyma in a suitable longitudinal plane.If there are multiple lesions in one subject requiring a second dose, the subject will have the option to undergo a 2nd contrast-enhanced study 30-minutes after the initial contrast dose, per dosing instructions in the package insert.
  Other Names: Definity; Microbubble contrast agent
  Arms: Perflutren Lipid Microsphere (Healthy subjects); Perflutren Lipid Microsphere (patients with kidney lesions)

SUMMARY:
The purpose of this research study is to evaluate contrast-enhanced ultrasound for kidney malignancies.

DETAILED DESCRIPTION:
This is an investigator-initiated, prospective study designed to evaluate the accuracy of contrast-enhanced ultrasound (CEUS) with microbubble contrast agent (perflutren lipid; Definity®) to identify malignancy in patients with kidney disease, a known risk factor for kidney malignancy, in whom a conventional ultrasound (US) or other prior imaging shows an indeterminate or suspicious kidney lesion.

The primary objective of the study is to estimate the sensitivity of CEUS in diagnosing kidney malignancy in patients with a risk factor for kidney malignancy and compare it to the current gold standard test in this patient population. Secondary analysis will include more optimal contrast-enhanced imaging with computed tomography (CT) or magnetic resonance imaging (MRI) in a subset of patients who can receive these studies. The study outcome will lead to immediate clinical application in patients with chronic kidney disease. Given the cost-effectiveness and adverse event profile, it has excellent potential to become established as first line diagnostics in the general patient population as well.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for the present study, patients must meet the following criteria:

1. Able to provide written informed consent
2. Willing to comply with protocol requirements
3. At least 18 years of age
4. Have kidney disease, defined as either chronic kidney disease (CKD) II-V, determined by estimated glomerular filtration rate (GFR) of <90 and derived from serum creatinine measurements, or albuminuria/proteinuria, determined by albumin to creatinine ratio or protein to creatinine ratio of >30mg/gm within 3 months of recruitment, or on dialysis or having received a kidney transplant or have biopsy proven kidney disease. In these latter cases, blood and urine tests are not necessary.
5. Have at least one kidney lesion identified but incompletely characterized on a non-contrasted US, CT, or MR exam for which the patient's provider recommends follow-up studies or further evaluation with additional imaging test(s).

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded for enrollment:

1. Critically ill or medically unstable and whose critical course during the observation period would be unpredictable (e.g., chronic obstructive pulmonary disease (COPD) requiring oxygen)
2. Known hypersensitivity to sulfur hexafluoride or to any component of perflutren lipid (Definity®)
3. Right to left shunt, severe pulmonary hypertension (Pulmonary artery pressure >90mmHg), or adult respiratory distress syndrome
4. Active cardiac disease including any of the following:

   * Severe congestive heart failure (class IV in accordance with the classification of the New York Heart Association)
   * Unstable angina
   * Severe arrhythmia (i.e., ventricular tachycardia, flutter fibrillation; ventricular premature complexes occurring close to the preceding T-wave, multifocal complexes)
   * Myocardial infarction within 14 days prior to the date of proposed Definity® administration
   * Uncontrolled systemic hypertension (systolic blood pressure (BP)>180 mm Hg and/or diastolic BP>100 mm Hg despite optimal medical management)
5. Is in an intensive care setting
6. Has an unstable neurological disease (e.g., cerebrovascular accident (including transient ischemic attacks (TIAs) within the 3 months before signing of informed consent
7. Has undergone an invasive procedure on kidney lesion (e.g., tissue biopsy, surgery, nonsurgical cytoreductive procedure) since identification of lesion via US without contrast
8. Has any other medical condition or other circumstances that would significantly decrease the chances of obtaining reliable data or of achieving the study objectives such as:

   * Mental illness
   * Drug abuse
9. Female patient who is pregnant or lactating (the possibility of pregnancy has to be excluded by negative point of care (POC), serum or urine beta-human chorionic gonadotropin (Β-HCG) results, obtained within 24 hours before the perflutren lipid administration, or on the basis of patient history, e.g., tubal ligation, hysterectomy or a minimum of 1 year without menses)
10. Obesity that limits obtainment of acceptable images

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-08-28 (Actual); Primary Completion 2021-03-19 (Actual); Study Completion 2021-03-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily Chang, M.D., Principal Investigator — University of North Carolina Kidney Center 7024 Burnette Womack CB#7155 Chapel Hill,NC 27599-7155
Locations (1):
- University of North Carolina of Chapel hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The controls without interaction were to be patients that declined enrollment who were willing to participate as controls. No participants agreed to participate in this arm.
Period: Overall Study
Arm/Group | Perflutren Lipid Microsphere (Healthy Subjects) | Perflutren Lipid Microsphere (Patients With Kidney Lesions) | Controls: No Interaction
Started | 5 | 20 | 0
Completed | 5 | 20 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The controls without interaction were to be patients that declined enrollment who were willing to participate as controls. No participants agreed to participate in this arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Perflutren Lipid Microsphere (Healthy Subjects) | Perflutren Lipid Microsphere (Patients With Kidney Lesions) | Controls: No Interaction | Total
Number analyzed (Participants) | 5 | 20 | 0 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 |  | 0
  Between 18 and 65 years | 5 | 15 |  | 20
  >=65 years | 0 | 5 |  | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (15) | 58 (11) |  | 56 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 |  | 8
  Male | 3 | 14 |  | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 |  | 1
  Not Hispanic or Latino | 5 | 18 |  | 23
  Unknown or Not Reported | 0 | 1 |  | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 |  | 0
  Asian | 0 | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 |  | 0
  Black or African American | 1 | 10 |  | 11
  White | 3 | 10 |  | 13
  More than one race | 0 | 0 |  | 0
  Unknown or Not Reported | 1 | 0 |  | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 20 |  | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Change in Radiologist's Lesion Evaluation
Description: Lesions will be assessed for change in size, calcification, and septation using Bosniak criteria to determine whether a lesion has progressed, regressed or is stable.
Time Frame: 1 year
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Perflutren Lipid Microsphere (Healthy Subjects) | Perflutren Lipid Microsphere (Patients With Kidney Lesions) | Controls: No Interaction
Number analyzed (Participants) | 5 | 20 | 0
Participants
  Stable | 0 | 11 |
  Progression | 0 | 1 |
  Regression | 0 | 2 |
  Unable to assess | 0 | 1 |
  Not applicable | 5 | 5 |

ADVERSE EVENTS:
Time Frame: 1 year following contrast administration
Description: The controls without interaction were to be patients that declined enrollment who were willing to participate as controls. No participants agreed to participate in this arm.
Arm/Group | Perflutren Lipid Microsphere (Healthy Subjects) | Perflutren Lipid Microsphere (Patients With Kidney Lesions) | Controls: No Interaction
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/20 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/20 | 0/0
Other Adverse Events (participants affected / at risk) | 0/5 | 0/20 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-02): https://cdn.clinicaltrials.gov/large-docs/76/NCT03196076/Prot_SAP_000.pdf